CLINICAL TRIAL: NCT03342989
Title: Speed of Processing Training for Cognitive Deficits After Delirium in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment not sufficient to justify continuation
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Richard Kennedy, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-300000471; R21AG057982-01 (NIH)
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Delirium; Dementia
Keywords: delirium; speed of processing; cognitive decline
MeSH Terms: conditions — Delirium; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speed of Processing Training (Experimental): Training involves detection, localization, and discrimination of briefly displayed stimuli (17-500 milliseconds) using tasks with varying demands on visual attention. Cognitive processing speed is defined as response accuracy at a given display duration, regardless of motor speed. Training involves detection, localization, and discrimination of briefly displayed stimuli (17-500 milliseconds) using tasks with varying demands on visual attention. Speed of processing is defined as response accuracy at a given display duration, regardless of motor speed. Training consists of 10 lab-based sessions over 5 weeks, followed by home-based practice on a tablet computer for 24 months with supportive home visits.
  Interventions: Behavioral: Speed of Processing Training
- Internet-Based Contact Control (Active Comparator): Training involves mentally stimulating activity and consists of three levels: (1) using a computer (e.g., mouse training, pull-down menus, selecting options), (2) internet search engine training, and (3) search engine proficiency tasks. Training consists of 10 lab-based sessions over 5 weeks, followed by home-based practice on a tablet computer for 24 months with supportive home visits.
  Interventions: Behavioral: Internet-Based Contact Control

INTERVENTIONS:
Behavioral: Speed of Processing Training — This intervention is based on computer-administered tasks that are used to evaluate Useful Field of View test, which measures discrimination between visually presented stimuli in the presence of distractors
  Arms: Speed of Processing Training
Behavioral: Internet-Based Contact Control — This intervention provides social contact and mentally stimulating activities that do not target speed of processing
  Arms: Internet-Based Contact Control

SUMMARY:
In this proposal, we will examine processing speed training (PST) as a potential intervention to reduce the risk of developing long-term cognitive impairment after a delirium episode.

DETAILED DESCRIPTION:
The overall goal of this project is to measure longitudinal cognitive function among hospitalized older adults after an episode of delirium, and examine an intervention (processing speed training, or PST) to slow the rate of cognitive decline that occurs after an episode of delirium compared to an Internet-based control condition (INT). We will initially recruit a cohort of 136 subjects who have experienced delirium, provide PST or INT training to them, and assess them on measures of cognition and instrumental activities of daily living (IADLs) after training and every 6 months thereafter for 24 to 36 months. We will perform a preliminary determination of the efficacy of PST after these 136 subjects have completed training, testing whether subjects receiving PST have better cognitive test scores immediately after training compared to subjects receiving INT. Assuming this preliminary test of efficacy shows short-term benefits for PST, we will recruit an additional 280 subjects who have experienced delirium and provide PST training to them. We will follow all 416 subjects for 24 to 36 months after their delirium episode to test whether subjects receiving PST have slower rates of decline over time compared to subjects receiving INT on measures of cognition and IADLs. A more detailed timeline of study procedures follows.

In Hospital (Month 0): We will initially identify subjects with delirium from the inpatient medical units at UAB Hospital. As part of UAB's Virtual ACE quality improvement project, nurses on the medical units administer the Nursing Delirium Screening Scale (NUDESC) to screen for delirium in all patients age ≥ 65 on admission and once per shift thereafter. After obtaining informed consent, we will collect a range of measures from the subject and family to make the diagnosis of delirium and rate its severity, as well as measures examining comorbidities potentially contributing to delirium. These measures for assessing delirium will be

* the NUDESC ratings from the medical record;
* the Confusion Assessment Method (CAM), a standard clinician-rated instrument for the diagnosis of delirium;
* the Delirium Symptom Interview (DSI), an interview administered by a clinician to standardize the assessment of delirium symptoms for rating the CAM;
* the Cognitive Test for Delirium (CTD), a general measure of cognition used to standardize the assessment of cognitive symptoms for rating the CAM;
* the Family Confusion Assessment Method (FAMCAM), which assesses the family's observation of symptoms of delirium (although this will not be required for delirium diagnosis);
* the chart-based review method for delirium (CHART-DEL), which collects information from the medical records about signs and symptoms that can indicate delirium;
* the Delirium Etiology Rating Checklist (DERC), a clinician-rated instrument that categorizes the different potential causes of delirium for the subject, based on information in the medical record on other medical conditions, current medications, neuroimaging (CT or MRI, if available), abnormal laboratory values (complete blood count, serum electrolytes and chemistries, liver function tests, and urine drug screen, if available);
* the Anticholinergic Burden Scale (ABS), which rates the contribution of the subject's medications to their episode of delirium.

Additional measures collected on comorbidities and factors affecting delirium will be

* demographics (age, race, gender);
* the AD8 and the Modified Blessed Dementia Rating Scale, which assess the family's observations of symptoms of dementia that preceded the episode of delirium;
* the Charlson Comorbidity Index (CCI), which assesses the presence of other medical conditions beyond delirium.

After the initial in-hospital assessment, we will continue to follow the subject for the remainder of their stay, using the CAM and the DRS-R-98 to monitor the duration of delirium. We will also collect the NUDESC assessments given by nursing staff on a daily basis.

Outpatient Baseline (Approximately Month 1, depending on length of hospitalization): Approximately 2 weeks after hospital discharge, we will contact subjects by telephone for follow-up. We will review the study procedures with the subject and use the CAM to see if their delirium has resolved. Once a subject's delirium has resolved, we will bring them to our offices for a comprehensive baseline assessment. Measures for this visit will examine cognition (particularly memory and executive function) and function (particularly activities of daily living and instrumental activities of daily living), as well as general health and mental health. Specific measures will be

* the CAM;
* the FAMCAM;
* the CTD;
* the AD8;
* the Wechsler Test of Adult Reading (WTAR), a vocabulary test to estimate IQ;
* the General Cognitive Performance (GCP) battery, a composite of the following neuropsychological tests

  * the Visual Search and Attention Test, measuring executive function and visuospatial skills;
  * the Hopkins Verbal Learning Test-Revised, measuring verbal memory;
  * the WAIS Digit Span Forward and Backward, measuring attention;
  * Category Fluency, measuring executive function and language;
  * Phonemic Fluency, measuring executive function and language;
  * the Boston Naming Test, measuring naming and language;
  * the RBANS Digit Symbol Test, measuring executive function and visuospatial skills;
  * the DKEFS Trail Making Test, measuring executive function and visuospatial skills;
* the Katz Activities of Daily Living (ADLs), which rates ability to perform basic activities for daily life;
* the Lawton Instrumental Activities of Daily Living (IADLs), which rates ability to perform more complex activities for daily life;
* the Timed IADLs, which measures speed at performing complex activities of daily life;
* the Geriatric Depression Scale (GDS), a standard measure of depressive symptoms in older adults;
* the Medical Outcomes Study 12-item Short Form (SF-12), a standard measure of overall health and quality of life;
* healthcare utilization (rehospitalization or institutionalization) since discharge.

PST or INT Training (Months 1 and 2): After the baseline assessment, we will randomize each subject to 10 sessions of PST or INT, which will be conducted in the outpatient setting at UAB for standardization. The PST training consists of computer-administered sessions in which a subject practices detection and discrimination of targets displayed for short periods of time. The INT training consists of sessions in which a subject practices general computer skills and use of Internet search engines.

Post-Training Assessment (Month 2): After lab-based training, subjects will complete a follow-up assessment that will repeat measures of cognition, function, and general health

* the GCP (neuropsychological testing);
* the Katz ADLs (functional status);
* the Lawton IADLs (functional status);
* the Timed IADLs (functional status);
* the GDS (mental health);
* the SF-12 (general health);
* the AD8 (dementia symptoms);
* healthcare utilization (rehosopitalization or institutionalization) since baseline.

Semiannual Assessments (Months 6, 12, 18, 24, 30, and 36): Subjects will continue to practice PST or INT at home with study-distributed tablet computers and supportive visits for the remainder of the study. Every 6 months, we will repeat measures of cognition, function, and general health

* the GCP (neuropsychological testing);
* the Katz ADLs (functional status);
* the Lawton IADLs (functional status);
* the Timed IADLs (functional status);
* the GDS (mental health);
* the SF-12 (general health);
* the AD8 (dementia symptoms AD8);
* healthcare utilization (rehospitalization or institutionalization) since previous visit;
* incident dementia.

For the determination of incident dementia, data on subjects scoring more than 1 standard deviation below the mean on 2 or more neuropsychological tests will be reviewed by a Clinical Consensus Panel, who will assign a diagnosis of mild cognitive impairment or dementia (if warranted) according to National Institute on Aging-Alzheimer's Association criteria.

Preliminary Evaluation of Short-Term Treatment Efficacy This evaluation will be examine short-term differences between groups on cognition (GCP) and function (Timed IADLs) at 2 months, after all 136 subjects have completed lab-based PST or INT training. We will also evaluate the effects of pre-existing cognitive impairment by comparing the effects of PST to those without pre-existing cognitive impairment. Using ANOVA to compare treatment groups, a sample size of N=136 will have greater than 80% power to detect a 30% difference in scores on the GCP, which is smaller than the 30% difference considered meaningful in trials for interventions in prodromal Alzheimer's disease. A sample size of N=136 will also be sufficient to allow comparisons between subjects with and without pre-existing cognitive impairment.

Recruitment of the Second Cohort Assuming the preliminary evaluation of treatment efficacy demonstrates positive effects for PST, we recruit 280 additional subjects while continuing to follow the original cohort of 136 subjects, so that our total cohort of 416 subjects will provide sufficient power to examine the effect of PST on cognitive and functional declines over time. Enrollment procedures and assessments for new subjects will be identical to those for the original cohort. After completion of PST or INT training, all subjects will be followed for 24 to 36 months (depending on the time of enrollment), with assessments every 6 months as described above.

Evaluation of Long-Term Treatment Efficacy We will evaluate efficacy by examining differences in the slope, or rate of change, on cognition (the GCP) and function (Timed IADLs) between the PST and INT groups over the follow-up period. We will also evaluate whether effects of PST on cognitive outcomes differs subjects with pre-existing MCI or mild dementia compared to those without pre-existing cognitive impairment. Using mixed effects models to compare slopes, a sample size of N=416 will have greater than 80% power to detect a difference between treatment groups. This will also be sufficient to allow comparisons between subjects with and without pre-existing cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* English speaking (English need not be first language);
* admission to the inpatient medical wards at University of Alabama at Birmingham Hospital;
* positive screen for delirium, defined as a score ≥ 1 on the Nursing Delirium Screening Scale, during hospitalization;
* presence of delirium, defined using the Confusion Assessment Method, during hospitalization;
* informant-rated AD8 score ≤ 6;
* living within 40 miles of the Birmingham, Alabama metro area.

Exclusion Criteria:

* active delirium at the time of baseline assessment after hospital discharge, defined using the Confusion Assessment Method;
* hospitalization in the previous 3 months prior to the index hospitalization;
* terminal condition with life expectancy < 6 months;
* inability to perform cognitive tests due to poor vision or hearing at baseline assessment;
* history of schizophrenia or other psychotic disorder;
* alcohol withdrawal delirium during hospitalization, history of alcohol abuse, or history of alcohol withdrawal in the previous 6 months;
* unable to provide informed consent at baseline visit (proxy consent may be used for in-hospital assessments).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
General Cognitive Performance Battery | 2 Month Follow-up
  Composite Neuropsychological Test Battery
General Cognitive Performance Battery | 24 Month Follow-up
  Composite Neuropsychological Test Battery

SECONDARY OUTCOMES:
Timed Instrumental Activities of Daily Living | 2 Month Follow-up
  Time to complete everyday activities
Timed Instrumental Activities of Daily Living | 24 Month Follow-up
  Time to complete everyday activities
Incident Dementia | 2 Month Follow-Up
  Time to Development of Dementia by Consensus Conference
Incident Dementia | 24 Month Follow-Up
  Time to Development of Dementia by Consensus Conference

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Kennedy, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Given the current lack of treatments for the cognitive and functional complications of delirium, we anticipate that this data will be of great interest to other researchers, both for exploring additional hypotheses that were not part of this proposal and as pilot data for designing future trials of other interventions in delirium. Data to be shared will consist of demographic and medical data, cognitive assessment data, and data on daily functioning collected as part of the study. Data will be stripped of personal identifiers prior to distribution. Data will be made available by request through a secure file-sharing service hosted by the University of Alabama at Birmingham (e.g., UAB Box). Interview data will be made available in file formats for a variety of statistical software (e.g., SPSS, SAS, R). All investigators will provide instructions on how to access the data in any publications and presentations utilizing data from this proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Access to the data by other investigators, and dissemination of information on how to access the data, will begin as soon as possible but no later than within one year of the completion of the funded project period for the parent award or upon acceptance of the data for publication, whichever is earlier.
Access Criteria: Data sets will be distributed to researchers at other institutions after approval by the study investigators. Researchers will be required to submit a data use agreement and a brief research proposal outlining the goals of the research and the specific data elements requested. All requests will also require IRB approval (or documentation of exemption from IRB review) by the researcher's institution prior to release as well as the UAB IRB.

REFERENCES:
- [Background] Wadley VG, Benz RL, Ball KK, Roenker DL, Edwards JD, Vance DE. Development and evaluation of home-based speed-of-processing training for older adults. Arch Phys Med Rehabil. 2006 Jun;87(6):757-63. doi: 10.1016/j.apmr.2006.02.027. PMID 16731209
- [Background] Inouye SK, Marcantonio ER, Kosar CM, Tommet D, Schmitt EM, Travison TG, Saczynski JS, Ngo LH, Alsop DC, Jones RN. The short-term and long-term relationship between delirium and cognitive trajectory in older surgical patients. Alzheimers Dement. 2016 Jul;12(7):766-75. doi: 10.1016/j.jalz.2016.03.005. Epub 2016 Apr 18. PMID 27103261